CLINICAL TRIAL: NCT05209906
Title: An Observation Study to Assess the Efficacy and Safety of Proportional Doses of Painkyl® in Patients With Breakthrough Cancer Pain
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Shing Leu, Head of Otorhinolaryngology Department (ENT), Mackay Memorial Hospital
Other Study IDs: 19MMHIS032e
Record Dates: First submitted 2021-12-24; First posted 2022-01-27 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fentanyl Buccal Soluble Film — Eligible patients will receive Painkyl® for dose of 200, 400, 600, 800, 1000 or 1200 mcg for the treatment of breakthrough pain according to around-the-clock morphine daily dose.

SUMMARY:
An open-label, single arm, observation study, to assess the efficacy and safety of proportional doses of Painkyl® in patients with breakthrough cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. cancer patients regularly experienced 1 to 3 breakthrough pain episodes per day that required additional opioids from pain control;
2. a current regimen of opioids equivalent to 60-360 mg/day of oral morphine or 25-150 mcg/hr of transdermal fentanyl for one week or longer;
3. at least partial relief of breakthrough pain by use of opioid therapy;
4. able to self-administer the study medication correctly or has an available adult caregiver to administer the study medication correctly;
5. willing and able to complete patient diary with each pain episode.
6. 20 to 80 years of age;

Exclusion Criteria:

1. rapidly escalating pain (e.g., regularly more than 3 breakthrough pain episodes per day) that are hard to be controlled by analgesics;
2. history of hypersensitivity or intolerance to fentanyl;
3. cardiopulmonary disease that, in the opinion of the investigator, would significantly increase the risk of respiratory depression;
4. psychiatric/cognitive or neurological impairment that would limit the subject's ability to understand or complete the diary;
5. Severe (Grade 4) mucositis (subjects with less than severe mucositis are permitted and must be instructed to not apply the Painkyl® film at a site of inflammation);
6. abnormal oral mucosa which will impede drug absorption;
7. recent history or current evidence of alcohol or other drug substance (licit or illicit) abuse;
8. use of an investigational drug or other rapid-onset opioids drugs within 4 weeks preceding this study;
9. pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients experienced breakthrough pain even under around-the-clock narcotic drug treatment.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients requiring dose titration | At study end (at least 30 subjects completed 2 doses of study treatment without dose titration), around 4 years
  Percentage of patients requiring dose titration

SECONDARY OUTCOMES:
Pain intensity changes at 5, 10, 15, 30 minutes after dosing | At study end (at least 30 subjects completed 2 doses of study treatment without dose titration), around 4 years
  Pain score at 5, 10, 15, 30 minutes after dosing vs. pain score before dosing. Pain scale (0-10, 0=no pain to 10=worst pain) will be recorded by subject at the time point of before Painkyl dosing, and at 5, 10, 15, 30 minutes after dosing.
Subjects' satisfaction | At study end (at least 30 subjects completed 2 doses of study treatment without dose titration), around 4 years
  Subjects' satisfaction (poor, fair, good, very good, excellent) will be recorded by subject for at least 2 assessment

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Chiang YH, Lien CT, Su WH, Yen TY, Chen YJ, Lai YL, Lim KH, Dai KY, Chung HP, Hung CY, Leu YS. Effectiveness of fentanyl buccal soluble film in cancer patients with inadequate breakthrough pain control. BMC Palliat Care. 2024 Jun 14;23(1):150. doi: 10.1186/s12904-024-01483-7. PMID 38877477